CLINICAL TRIAL: NCT01828216
Title: A Randomized Controlled Study Assessing the Role of an Ambulatory Approach Versus the Conventional Approach in Managing Suspected Obstructive Sleep Apnoea Syndrome
Brief Title: Ambulatory Versus Conventional Approach Diagnosing OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: amb_hosp_OSA
Record Dates: First submitted 2013-04-08; First posted 2013-04-10 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-02

CONDITIONS: OSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional polysomnography (Active Comparator): Conventional PSG will be performed as in-patient at Prince of Wales Hospital for every subject in this group, recording electroencephalogram, electro-oculogram, submental electromyogram, bilateral anterior tibial electromyogram, electrocardiogram, chest & abdominal wall movement by inductance plethysmography, airflow measured by a nasal pressure transducer & supplemented by oronasal airflow thermistor, & finger pulse oximetry.
  Interventions: Device: conventional polysomnography
- Home sleep study (Active Comparator): The home sleep study is a pocket-sized digital recording device. It is a multi-channel screening tool that measures airflow through a nasal cannula connected to a pressure transducer, providing an apnea-hypopnea index (AHI) based on recording time. It also detects both respiratory and abdominal efforts through the effort sensor and can differentiate between obstructive and central events.
  Interventions: Device: Home sleep study

INTERVENTIONS:
Device: Home sleep study — The home sleep study is a pocket-sized digital recording device. It is a multi-channel screening tool that measures airflow through a nasal cannula connected to a pressure transducer, providing an apnea-hypopnea index (AHI) based on recording time. It also detects both respiratory and abdominal efforts through the effort sensor and can differentiate between obstructive and central events
  Arms: Home sleep study
Device: conventional polysomnography — conventional type I sleep study according to international guidelines
  Arms: Conventional polysomnography

SUMMARY:
Very few studies have examined different models of care involving initial ambulatory home-based diagnosis in diagnosing obstructive sleep apnea (OSA), identifying patients who benefit from continuous positive airway pressure (CPAP), and reducing the need for polysomnography (PSG). This study aims to assess the role of an ambulatory approach with home diagnostic sleep study. We hypothesize that the ambulatory approach is as good as the conventional approach in managing OSA in terms of improvement of clinical outcome but the former approach will lead to substantial cost savings.

DETAILED DESCRIPTION:
We conducted a prospective, randomized, controlled continuous positive airway pressure (CPAP) parallel study on new referrals to the Respiratory Clinic, Prince of Wales Hospital, with suspected obstructive sleep apnea (OSAS). OSAS was defined by apnea-hypopnea index(AHI) 5/hr or more of sleep plus excessive daytime sleepiness or two of the following symptoms: choking or gasping during sleep, recurrent awakenings from sleep, unrefreshed sleep, daytime fatigue, and impaired concentration. All patients with suspected OSAS underwent assessment at the clinic with the Epworth sleepiness score(ESS) and symptoms evaluation. Patients who had ESS score>9 or at least two OSAS symptoms as described above were invited to join the study. They were randomized into either group A)home-based management approach or group B)hospital-based management approach by a random table by a third party not involved in the trial.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of OSA with home sleep study AHI >= 15/hr.

Exclusion Criteria:

* unstable cardiovascular diseases (e.g. recent unstable angina, myocardial infarction, stroke or transient ischemic attack within the previous 6 months or severe left ventricular failure)
* neuromuscular disease affecting or potentially affecting respiratory muscles
* moderate to severe respiratory disease (i.e. breathlessness affecting activities of daily living) or documented hypoxemia or awake oxygen saturation of <92%
* psychiatric disease that limits the ability to give informed consent or complete the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong SAR, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ng SS, Tam W, Chan TO, To KW, Ngai J, Chan KKP, Yip WH, Lo RL, Yiu K, Ko FW, Hui DS. Use of Berlin questionnaire in comparison to polysomnography and home sleep study in patients with obstructive sleep apnea. Respir Res. 2019 Feb 22;20(1):40. doi: 10.1186/s12931-019-1009-y. PMID 30795760

RESULTS

PARTICIPANT FLOW:
Groups:
- In-hospital Sleep Study: Conventional polysomnography will be performed as in-patient at Prince of Wales Hospital for every subject in this group, recording electroencephalogram, electro-oculogram, submental electromyogram, bilateral anterior tibial electromyogram, electrocardiogram, chest & abdominal wall movement by inductance plethysmography, airflow measured by a nasal pressure transducer & supplemented by oronasal airflow thermistor, & finger pulse oximetry.
- Ambulatory Sleep Study: The home sleep study is a pocket-sized digital recording device. It is a multi-channel screening tool that measures airflow through a nasal cannula connected to a pressure transducer, providing an apnea-hypopnea index (AHI) based on recording time. It also detects both respiratory and abdominal efforts through the effort sensor and can differentiate between obstructive and central events.
Period: Overall Study
Arm/Group | In-hospital Sleep Study | Ambulatory Sleep Study
Started | 159 | 157
Completed | 159 | 157
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ambulatory Sleep Study: home sleep study is a pocket-sized digital recording device. It is a multi-channel screening tool that measures airflow through a nasal cannula connected to a pressure transducer, providing an apnea-hypopnea index (AHI) based on recording time. It also detects both respiratory and abdominal efforts through the effort sensor and can differentiate between obstructive and central events.
- Total: Total of all reporting groups
Arm/Group | In-hospital Sleep Study | Ambulatory Sleep Study | Total
Number analyzed (Participants) | 159 | 157 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (11.3) | 51 (12.9) | 51.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 50 | 91
  Male | 118 | 107 | 225

OUTCOME MEASURES:

1. Primary Outcome: Change in Epworth Sleepiness Score (ESS) Before and After 3 Months of Continuous Positive Airway Pressure (CPAP) Treatment
Description: The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness that is measured by use of a very short questionnaire. The questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 to 3 for eight different situations that most people engage in during their daily lives, though not necessarily every day. The scores for the eight questions are added together to obtain a single number. A number in the 0-9 range is considered to be normal while a number in the 10-24 range indicates that expert medical advice should be sought.
Time Frame: Baseline and 3 months
Population: Following detection of apnea-hypopnea index (AHI) of 15 events per hour or more by home sleep study or polysomnography, patients received CPAP therapy for 3 months after an overnight autoCPAP titration at in-hospital or ambulatory home setting.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- In-hospital CPAP Titration; Ambulatory CPAP Titration: Following detection of apnea-hypopnea index (AHI) of 15 events per hour or more by home sleep study or polysomnography, patients received CPAP therapy for 3 months after an overnight autoCPAP titration at in-hospital or ambulatory home setting.
Arm/Group | In-hospital CPAP Titration | Ambulatory CPAP Titration
Number analyzed (Participants) | 86 | 86
units on a scale | -2.2 (5.2) | -3.5 (5.0)

2. Secondary Outcome: Difference in Healthcare Costs Between Ambulatory and Hospital Approach
Time Frame: within 24 months
Measure: Mean (Standard Deviation); unit: Hong Kong Dollars
Arm/Group | In-hospital Sleep Study | Ambulatory Sleep Study
Number analyzed (Participants) | 69 | 62
Hong Kong Dollars | 16178 (2288) | 2332 (944)

ADVERSE EVENTS:
Arm/Group | In-hospital Sleep Study | Ambulatory Sleep Study
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/157
Other Adverse Events (participants affected / at risk) | 0/159 | 0/157

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No